CLINICAL TRIAL: NCT01936740
Title: Comparison of Two Phacoemulsification-methods: HF EasyTip 2.2mm vs. HF EasyTip 2.8mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Ao.Univ.-Prof. Dr.med.univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Ek Nr: 1268/2012
Record Dates: First submitted 2013-09-03; First posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Cataracts
Keywords: Efficacy and Safety
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- HF easyTip 2.2mm (Other): The phacoemulsifications tip used was the easyTip 2.2mm tip (Oertli Instruments, Berneck, Switzerland). The cristaline lens was divided into four quadrants using an aspiration flow rate of 10ml/min and vacuum of 70 mmHg. The quadrants were aspirated using the following linear power and fluidic settings: aspiration flow rate 45ml/min, vacuum 600 mmHg, bottle height 100cm.
  Interventions: Procedure: cataract surgery
- HF easyTip 2.8mm (Other): The phacoemulsifications tip used was the easyTip 2.8mm tip (Oertli Instruments, Berneck, Switzerland). The cristaline lens was divided into four quadrants using an aspiration flow rate of 10ml/min and vacuum of 70 mmHg. The quadrants were aspirated using the following linear power and fluidic settings: aspiration flow rate 50ml/min, vacuum 600 mmHg, bottle height 100cm.
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery

SUMMARY:
The aim of this study was to compare the intraoperative efficiency, safety and postoperative outcomes of cataract surgery with two different "high-fluidic" settings.

ELIGIBILITY:
Inclusion Criteria:

* bilateral age-related cataract
* good overall physical constitution
* LOCS 2-5

Exclusion Criteria:

* previous intraocular surgery or ocular trauma
* previous corneal pathology
* previous endothelial cell count <1200
* glaucoma
* uveitis
* PEX
* diabetic retinopathy and any other severe retinal pathology that would make a postoperative visual acuity of 20/40 (decimal equivalent = 0.5) or better unlikely
* intraocular complication like posterior capsular
* postoperative comlpications (e.g. postoperative uveitis)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
phacoemulsification time | intraoperative
  time spent for the phacoemulsification process was the phacoemulsification tip time (PTT) needed to divide the nucleus and the PTT needed to conquer it
effective phacoemulsification time | intraoperative
  time in seconds required had 100% power been used throughout the phacoemulsification process documented for the separation of the nucleus (divide) and the aspiration of the quadrants (conquer)
fluid volume | intraoperative
  amount of BSS used for dividing and conquering

SECONDARY OUTCOMES:
postoperative corneal oedema | 1 day, 1 week, 6 months
  central corneal thickness
postoperative endotheial cell loss | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology and Optometry of the Medical University Vienna, Vienna, Vienna, Austria